CLINICAL TRIAL: NCT04697420
Title: Transversus Abdominis Plane Block Versus Paravertebral Block for Post-operative Pain Relief Following Open Renal Surgeries: a Randomized Clinical Trial
Brief Title: Transversus Abdominis Plane Block Versus Paravertebral Block for Post Operative Pain Relief in Open Renal Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Hussein Ali, Resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AHAAssiut
Record Dates: First submitted 2020-12-29; First posted 2021-01-06 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (P) (Experimental): the patients were received paravertebral block to control pain postoperatively.
  Interventions: Procedure: Thoracic paravertebral block
- Group (T) (Experimental): the patients were received transversus abdomins plane (TAP) block to control pain postoperatively.
  Interventions: Procedure: Transversus abdominis plane block

INTERVENTIONS:
Procedure: Thoracic paravertebral block — Thoracic paravertebral block is a technique in which , the local anesthetic agent is injected in the paravertebral space to anesthetise the spinal nerves after emerging from the vertebral canal in order to provide analgesia in the thoracic and upper abdominal area .
  Arms: Group (P)
Procedure: Transversus abdominis plane block — Transversus abdominis plane block is a technique is mostly done under ultrasound guidance to identify the transversus plane between the internal oblique muscle and the transverses abdominis muscle , the space in which the neurovascular supply of the anterior abdominal wall is present , and hence the injection of local anesthetic agent in this space results in anesthesia of the anterolateral aspect of the abdominal wall.
  Arms: Group (T)

SUMMARY:
Pain relief after renal surgeries is essential as it may lead to reduction in the incidence of many post operative complications .

There are a lot of regional anesthetic techniques to provide analgesia postoperatively as paravertebral block (PVB) and transversus abdominis plane (TAP) block.

TAP block has been used to provide postoperative analgesia in a lot of abdominal surgeries including upper abdominal surgeries.It is safer technique than PVB, but the effectiveness of TAP block is unknown in comparison with PVB in post operative analgesia after renal surgeries .

DETAILED DESCRIPTION:
Pain relief after renal surgeries is essential as it may lead to reduction in the incidence of post operative respiratory complications . A lot of patients presented to these operations may have comorbidities as impaired renal function and respiratory problems , conditions like these may contraindicate aministration of systemic analgesia as opioids .

There are a lot of techniques to provide analgesia postoperatively as paravertebral block (PVB) and transversus abdominis plane (TAP) block .

Paravertebral block is effective technique for post operative analgesia for upper abdominal surgeries , but it may be associated with some complications as : pneumothorax , spread of local anesthetic to the epidural space and paravertebral blood vessels , and this may lead to systemic toxicity of local anesthetic .

TAP block has been used to provide postoperative analgesia in a lot of abdominal surgeries including upper abdominal surgeries , but it is safer technique than PVB , but the effectiveness of TAP block is unknown in comparison with PVB in post operative analgesia after renal surgeries .

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 60 years
* ASA I-II class

Exclusion Criteria:

* Patient refusal
* Any contraindication of regional anesthesia block (Coagulopathy,infection at the needle insertion site)
* Patients with allergy to amide local anesthetics or medication included in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
comparison between the post operative analgesic effect of transversus abdominis plane block and paravertebral block | 24 hours
  comparison between the post operative analgesic effect of transversus abdominis plane block and paravertebral block by the following assessment methods: Visual Analogue Scale score (VAS) immediately postoperative and through the first 24 hours postoperativly, total analgesic consumption through the first 24 hours postoperatively, and time of first analgesic request in the postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Essam Ezzat, Professor, Study Director — Professor of anesthesia, intensive care and pain management , formerly head of the department
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No